CLINICAL TRIAL: NCT02102724
Title: Fish Oil for HIV-Related Inflamm-aging and Immune Senescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5P20MD006886 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: HIV Infection
Keywords: African Americans; Older Adults
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two arms:
  Intervention arm = fish oil Control arm = placebo.
Who Masked: Participant, Investigator
Masking Description: All gelcaps were overencapsulated to mask their contents
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish Oil (Experimental): Participants will receive fish oil gelcaps that contain 1.6 grams of omega-3 fatty acids (800 mg of EPA, 600 mg DHA, 200 mg other omega-3 fatty acids) for 12 weeks.
  Interventions: Dietary Supplement: Fish oil that contains omega-3 fatty acids
- Placebo (Placebo Comparator): Participants will receive 1 gram of oleic sunflower oil for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish oil that contains omega-3 fatty acids — Fish oil gelcaps that contain 800 mg of EPA, 600 mg of DHA, 200 mg other omega-3 fatty acids
  Other Names: Carlson Brand fish oil
  Arms: Fish Oil
Dietary Supplement: Placebo — Gelcaps that contain 1 gram of oleic sunflower oil
  Arms: Placebo

SUMMARY:
HIV infection is associated with premature aging of the immune system. It is believe that the persistent inflammation that accompanies HIV infection is a major contributor to premature immune aging. Fish oil has well-documented anti-inflammatory properties. In this randomized, clinical trial, we're testing whether a 12-week course of fish oil supplementation will reverse premature aging in HIV-infected older adults.

DETAILED DESCRIPTION:
Due to treatment advances, the number of persons > 50 years old who are living with HIV/AIDS in the United States (US) has steadily increased. African Americans (AA) represent a disproportionate number of HIV/AIDS cases in this age group, with infection rates 12 times higher than among whites (51.7 per 100,000 compared to 4.2 per 100,000). Limited data suggest that older HIV+ AA are characterized by health status disparities. One cohort study of older, largely minority HIV+ persons (N=121, AA=83%;mean age=54), found that 34% had metabolic syndrome and 50% had a Framingham Cardiac Risk score > 10%. HIV+ older adults of all races show a premature onset of other age-associated co-morbidities, such as osteoporosis, non-AIDS malignancies, and cardiovascular disease (CVD). These co-morbidities have been linked to persistent inflammation and persistently elevated serum levels of proinflammatory cytokines that mimic an aging phenotype known as "inflamm-aging." In both middle-aged HIV+ persons and older HIV seronegative adults, inflamm-aging is associated with more limited T cell repertoires and increased risk for morbidities and mortality. In HIV infection, inflamm-aging is postulated to be maintained (a) by the constant antigen burden imposed by HIV and other chronic viral co-pathogens, such as cytomegalovirus (CMV), and (b) by HIV-induced disruption of intestinal epithelial integrity with subsequent translocation of gut microflora into the systemic circulation. Our hypothesis is that inflamm-aging is responsible for the premature immune senescence associated with HIV infection in aging individuals. Immune senescence, characterized by diminished replicative capacity, has been observed in middle-aged persons treated with highly active antiretroviral therapy (HAART) who achieve immune reconstitution and undetectable viral loads. Senescent cells are characterized by the absence of the surface marker CD28, and in advanced senescence express CD57 (CD28-/CD57+ phenotype). Because premature senescence leads to loss of anti-HIV cell-mediated immune responses and accelerated HIV disease progression,there is an urgent need to test new treatment strategies to reduce inflamm-aging and subsequent immune senescence.

Fish oil may be an effective treatment option for reducing HIV-related inflamm-aging. Cold water fish are rich in the omega-3 highly unsaturated fatty acids (HUFA) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), which have anti-inflammatory effects. When consumed as fish or fish oil supplements, EPA and DHA replace arachidonic acid in cell membranes and inhibit the synthesis of proinflammatory arachidonic acid metabolites, such as prostaglandins and leukotrienes. Moreover, animal and in vitro studies have shown that EPA and DHA stimulate regeneration of intestinal mucosa damaged by methotrexate,16 IL-4, and experimental ulcerative colitis. Yet, to date, no studies have been conducted on the effects of fish oil for reducing HIV-related inflamm-aging and reversing immune senescence.

The purpose of this study is to explore the safety and estimate the effect size of fish oil to modulate parameters of inflamm-aging and immune senescence in HIV+ older adults. Participants will receive either 1.6 grams of omega-3 fatty acids (800 mg of EPA, 600 mg DHA, 200 mg other omega-3 fatty acids) or placebo for 12 weeks. We expect to find a reduction in inflammatory markers and the percentage of CD8+ and CD4+ T lymphocytes that exhibit a senescent phenotype in the fish oil condition, but not in the control condition, at 12 weeks. We expect to find no difference between the conditions on the safety parameters at 4 and 12 weeks.

The specific aims are:

Aim 1. To assess the safety of the fish oil condition by comparing it to the control condition at 4 and 12 weeks, controlling for covariates (demographics, lifestyle, medications including HAART, fish oil supplement adherence, intercurrent illnesses), on

1. HIV disease parameters (CD4+ T cell counts and HIV RNA levels)
2. Drug toxicity (liver function tests and serum creatinine)
3. Adverse events (e.g., diarrhea, vomiting)

Aim 2. To estimate the effect size of the fish oil condition at 12 weeks, controlling for covariates, by comparing the following cell surface molecules and intracellular and soluble inflammatory markers before and after fish oil

1. Markers of immune senescence on CD8+ T lymphocytes: percentage of CD8+/CD28- T lymphocytes, a phenotype of immune senescence (primary outcome); percentage of CD8+/CD28-/CD57- T lymphocytes (an intermediate senescent phenotype); percentage of CD8+/CD28-/CD57+ T lymphocytes (a terminally differentiated senescent phenotype)
2. Markers of immune senescence on CD4+ T lymphocytes: percentage of CD4+/CD28- T lymphocytes; percentage of CD4+/CD28-/CD57- T lymphocytes; percentage of CD4+/CD28-/CD57+ T lymphocytes
3. Markers of inflammation: plasma hsCRP and intracellular concentrations of TNF-alpha, IL-6, and gamma IFN

Aim 3: To estimate the effect size of the fish oil condition at 12 weeks on gut permeability, controlling for covariates, by comparing the following indirect markers of gut permeability before and after fish oil

1. Endotoxin
2. Soluble mouse CD14
3. Endotoxin binding antibody
4. Lipopolysaccharide binding protein

ELIGIBILITY:
Inclusion Criteria:

* documented HIV infection
* between 40 and 70 years of age
* clinically stable HIV disease as evidenced by a CD4+ T lymphocyte count of > 250 cells/mm3
* platelet count between 150,000 and 400,000 cells/mm3 to reduce bleeding risks associated with omega 3-fatty acids
* treatment with a stable HAART regimen for at least six months prior to study entry
* plasma HIV RNA < 75 copies/ml for at least 12 months
* elevated plasma concentration of hsCRP (> 2.0 mg/L).

Exclusion Criteria:

* use within the past month of drugs (e.g., statins, steroids, hormones) and supplements (e.g., omega-3 fatty acids, glucosamine/chondroitin) that have anti-inflammatory effects (excluding non-regular use of aspirin or NSAIDS), or medications or supplements that affect bleeding (e.g., heparin, warfarin, clopidogrel, garlic, ginseng)
* allergy to fish or shellfish
* chronic inflammatory condition (e.g., asthma, rheumatoid arthritis), opportunistic infection or cancer, renal impairment (serum creatinine > 2.0 mg/dL), thrombocytopenia (platelet count < 150,000/mm3), bleeding episodes (e.g., gum bleeding, nosebleeds), or a metabolic condition (e.g., diabetes mellitus, thyroid disease)
* body mass index of > 35, since obesity is associated with inflammation
* impaired liver function as evidenced by liver enzyme elevations > three times the upper limit of normal (AST or ALT > 150 IU/L)
* history of prostate cancer
* LDL cholesterol level > 120 mg/dL
* lifestyle exclusion factors include use of illicit drugs and consumption of > 3 alcoholic drinks/day

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Swanson, PhD, RN, Principal Investigator — Rush University College of Nursing
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will receive 1 gram of oleic sunflower oil for 12 weeks.
  Fish oil that contains omega-3 fatty acids: Fish oil gelcaps that contain 800 mg of EPA, 600 mg of DHA, 200 mg other omega-3 fatty acids
Period: Overall Study
Arm/Group | Fish Oil | Placebo
Started | 18 | 19
Completed | 16 | 18
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — surgery for brain aneurysm | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (5.4) | 53 (6.1) | 54 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Markers of Immune Senescence Between Baseline Values and Values After 12 Weeks of Supplementation
Description: Markers of immune senescence will include change in the expression of the senescence markers CD28 and CD57 on the surface of peripheral CD4+ and CD8+ T lymphocytes. We will measure the percentage of CD4+ and CD8+ T lymphocytes that are CD28-/CD57- or CD28-/CD57+. We will subtract the percentage obtained at Week 12 from the baseline percentage to calculate the change scores.
Time Frame: End of 12-Week Supplementation Period
Population: Wilcoxon rank sum tests for intergroup change scores
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 18 | 19
percentage of cells
  Percent CD4+ cells CD28+/CD57- | 1.87 [-2.8 to 6.5] | 4.22 [-3.5 to 11.9]
  Percent CD4+ cells CD28-/CD57- | -2.83 [-6.9 to 1.2] | -1.56 [-3.0 to -0.08]
  Percent CD4+ cells CD28-/CD57+ | 0.69 [-1.2 to 2.5] | -2.41 [-9.6 to 4.8]
  Percent CD8+ cells CD28+/CD57- | -1.58 [-10.8 to 7.7] | -4.63 [-19.6 to 10.4]
  Percent CD8+ cells CD28-/CD57- | -3.6 [-7.7 to 0.5] | 0.79 [-4.8 to 6.4]
  Percent CD8+ cells CD28-/CD57+ | -2.37 [-8.7 to 4.4] | 1.96 [-6.2 to 10.1]
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; The null hypotheses were that there are no differences between the two groups' change scores for any study outcomes. The power analysis was based on a study of krill oil for reducing CRP levels in persons with arthritis (N = 90) that yielded an effect size (Cohen's d) of 1.2. A sample size of 37 was determined to yield a power of 0.80 to detect an effect size of 1.0 with a two-tailed alpha of 0.05; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); The change scores of the two groups (week 12 minus baseline) were compared using Wilcoxon rank sum tests

ADVERSE EVENTS:
Time Frame: Over the 12-week supplementation period
Description: Adverse event data were collected at baseline, week four and week 12.
Arm/Group | Fish Oil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/19
Other Adverse Events (participants affected / at risk) | 8/18 | 4/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil (N=18) | Placebo (N=19)
lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
brain aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil (N=18) | Placebo (N=19)
GI disturbance (Gastrointestinal disorders) | 8 (8) | 4 (4)

LIMITATIONS AND CAVEATS:
Small sample size; only single dose tested; duration may be too short to detect effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No